CLINICAL TRIAL: NCT04352699
Title: Outcomes of naïve Patients Operated on for an Urological Cancer or Emergency During Periods of Social COVID-19 Containment: is it Reasonable to Limit Access to Surgical Care for All?
Brief Title: Outcomes of Urological Surgery During Periods of Social COVID-19 Containemnt: is it Reasonable to Limit Access to Surgical Care for All?
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20urocovid01
Record Dates: First submitted 2020-04-14; First posted 2020-04-20 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-04

CONDITIONS: Surgery; Complication of Surgical Procedure; COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Naive patients: Group of naive patients who have undergone elective or emergency surgery during the study period

SUMMARY:
The French healthcare system has been strongly mobilized since the start of the Covid-19 epidemic to take care of patients with Covid-19. This should not overlook the fact that some treatments, surgeries and examinations of non-Covid-19 patients must imperatively be maintained according to the assessment of their risk-benefit balance. In context, it appears that this is not always the case. In addition to the necessary social containment measures, there are general limitations on patient access to the operating theater, neglecting the individual interest of naive non-Covid-19 patients. Certain studies which report a higher and earlier risk of death of undetected and ultimately operated Covid-19 patients has reinforced, as a precaution, the massive deprogramming of naive patients and the restrictive access of surgical care for all. We believe that this could lead to a risk of delayed treatments and renunciation of care for naive patients who should not be considered at risk a priori in the event of surgery. The individual clinical and local health context should be first considered for appropriate surgical decision-making.

As such, the French Department of Health and Human Services (DGS) has given general guidelines regarding the maintenance of follow-up and care for non-Covid-19 patients in this context of containment and major mobilization of health care professionals to care for people with COVID. Surgeries which could not be postponed because of the patient's status or if their postponement exposed to a significant risk of loss of chance, if needed in the light of the recommendations issued by learned societies, were concerned. In this sense, the investigator have selected the naive Covid-19 patients from Nice Hospital who should benefit from elective or urgent urological surgeries, taking into account their individual risk and the territorial epidemic rate. Their rate of ICU stays following their surgery has been analysed and their surgical follow-up outcomes during the epidemic period evaluated, according to the anti-Covid-19 measures established in Nice Hospital by comparing them to an earlier period without Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* naive patient for elective or emergency urological surgery

Exclusion Criteria:

* minor less than 18 year old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient selected for elective surgery or emergency surgery in the time frame
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of UCI admission for surgery-related complication | 1 month and a half
  Admission Rate is defined by the number of patient admitted to ICU due to surgical-related complication during 1 month and a half included in the Covid-19 period out of the number of operated patient in the same time within the institution

SECONDARY OUTCOMES:
Rate of surgery-specific death | 1 month and a half
  Number of patient dead from Covid after surgery out of number of dead patients in the same time frame within the institution
Rate of coronaviruse positive serologies | 1 month and a half
  Number of positives serologies within the cohort over a 1 month follow-up period. And coronaviruse related symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No
no data sharing plan has been established